CLINICAL TRIAL: NCT01265238
Title: Study of the Efficacy and Safety of the Neuro-orthopaedic Surgery in the Treatment of the Spastic Equinovarus Foot With ICF Assessment
Brief Title: Neuro-orthopaedic Surgery in the Treatment of the Spastic Equinovarus Foot
Status: Completed | Type: Observational
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Deltombe Thierry, Professeur Clinique, University Hospital of Mont-Godinne
Other Study IDs: MG-SEF-ICF-1
Record Dates: First submitted 2010-12-20; First posted 2010-12-23 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Spasticity; Spastic Foot; Stroke
Keywords: Spastic equinovarus foot; Stroke; Neurotomy; Tendon surgery
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Spastic equinovarus foot (SEF) is a major cause of disability in stroke patients. Treatments may include physical therapy, orthosis, botulinum toxin (BTX) injections, selective tibial neurotomy and tendon lengthening and/or transfer.

Until now, no study has been conducted to assess the result of neuro-orthopaedic surgery in the treatment of SEF.

The aim of this study is to evaluate the benefit of neuro-orthopaedic surgery (selective neurotomy and/or Achilles tendon lengthening and/or tibialis anterior transfer) in case of SEF according to the 3 domains of the International Classification of Functioning, Disability and Health (ICF)of the World Health organisation (WHO)

DETAILED DESCRIPTION:
INTRODUCTION

Stroke is the third cause of death and the leading cause of handicap among industrialized countries (1). Spasticity following stroke is responsible for spastic equinovarus foot (SEF) in 18% of cases (2). Spastic equinovarus foot is due to spasticity (muscle hypertonia) of the calf muscles (soleus, gastrocnemius and tibialis posterior), often complicated by contracture and by the weakness of peroneus longus and peroneus brevis muscles (3). Therefore, stroke patients walk slowly, and often require assistive device as orthosis or canes. This disability limits their social participation and their quality of life.

Spastic equinovarus foot treatments include oral medications, physical therapy, orthosis, chemical denervations (botulinum toxin, alcohol or phenol injections), selective neurotomy and orthopedic surgery (3). Selective neurotomy is a neurosurgical procedure consisting in partially and selectively cutting motor branches innervating the spastic muscles providing a permanent treatment of the spasticity (3). Orthopaedic surgery consists in Achilles tendon lengthening and tibialis anterior transfer (3). The efficacy of mixed neur-orthopaedic surgery has never been prospectively assess according to the ICF classification.

OBJECTIVES

The aim of the present project is to study the effectiveness of neuro-orthopaedic surgery (neurotomy and tendon surgery) in the treatment of SEF.

The functional assessment will explore the three ICF domains.

METHODS

The investigators will recruit 50 chronic spastic patients presenting with SEF. The surgical treatment will be decided according to the improvement obtained by an anaesthetic diagnostic tibial motor nerve branches block (5) followed by an interdisciplinary discussion.

Patients will be assessed before treatment, 2 months, 1 year and 2 years after treatment among the 3 ICF domains. Impairments will be assessed by the Stoke Impairment Assessment Set (SIAS), the Ashworth and Tardieu scales (spasticity) and the MRC scale (muscle strength). Gait disorders will be evaluated by a video analysis. Disability will be evaluated by the ABILOCO scale (6) and the participation (quality of life) by the SATIS-Stroke questionnaire (7) and the SF-36 questionnaire.

The patients selection, the lidocaine hyperselective diagnostic blocks, the selective neurotomy and the tendon surgery will be achieved by the medical doctors participants to the spasticity group. The functional assessment will be achieved by the physical therapists of the PMR department (blinded assessor).

PERSPECTIVE

The investigators hope to demonstrate the benefit of neuro-orthopaedic surgery in case of SEF according to the 3 domains of the ICF (8)

ELIGIBILITY:
Inclusion Criteria:

* central neurological disease lasting from more than 6 months
* spastic equinovarus foot due to spasticity and/or contracture
* patient able to walk barefoot
* insufficient benefit from physical therapy and/or orthosis

Exclusion Criteria:

* pregnant women
* botulinum toxin injection in the last 4 months
* previous surgery for SEF

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with central neurological disease (stroke, traumatic brain injury, spinal cord injury, multiple sclerosis) suffering from a spastic equinovarus foot referred to an interdisciplinary spasticity group in a University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Stroke impairment assessment scale, Ashworth scale, MRC scale, gait speed, Abiloco, SF36 and SATIS-stroke | Before treatment (T0)
  Scale measuring disability, incapacity and participation
Stroke impairment assessment scale, Ashworth scale, MRC scale, gait speed, Abiloco, SF36 and SATIS-stroke | 2 months after surgery (T1)
  Scales measuring disability, incapacity and participation
Stroke impairment assessment scale, Ashworth scale, MRC scale, gait speed, Abiloco, SF36 and SATIS-stroke | 1 year after surgery (T2)
  Scale measuring disability, incapacity and participation

CONTACTS AND LOCATIONS:
Overall Officials: Thierry M Deltombe, M.D., Principal Investigator — University Hospital of Mont-Godinne, Université Catholique de Louvain
Locations (1):
- University Hospital of Mont-Godinne, Yvoir, Belgium

REFERENCES:
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Recovery of walking function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 Jan;76(1):27-32. doi: 10.1016/s0003-9993(95)80038-7. PMID 7811170
- [Background] Verdie C, Daviet JC, Borie MJ, Popielarz S, Munoz M, Salle JY, Rebeyrotte I, Dudognon P. [Epidemiology of pes varus and/or equinus one year after a first cerebral hemisphere stroke: apropos of a cohort of 86 patients]. Ann Readapt Med Phys. 2004 Mar;47(2):81-6. doi: 10.1016/j.annrmp.2003.10.005. French. PMID 15013602
- [Background] Deltombe T, Gustin T. Selective tibial neurotomy in the treatment of spastic equinovarus foot in hemiplegic patients: a 2-year longitudinal follow-up of 30 cases. Arch Phys Med Rehabil. 2010 Jul;91(7):1025-30. doi: 10.1016/j.apmr.2010.04.010. PMID 20599040
- [Background] Deltombe T, De Wispelaere JF, Gustin T, Jamart J, Hanson P. Selective blocks of the motor nerve branches to the soleus and tibialis posterior muscles in the management of the spastic equinovarus foot. Arch Phys Med Rehabil. 2004 Jan;85(1):54-8. doi: 10.1016/s0003-9993(03)00405-2. PMID 14970968
- [Background] Caty GD, Arnould C, Stoquart GG, Thonnard JL, Lejeune TM. ABILOCO: a Rasch-built 13-item questionnaire to assess locomotion ability in stroke patients. Arch Phys Med Rehabil. 2008 Feb;89(2):284-90. doi: 10.1016/j.apmr.2007.08.155. PMID 18226652
- [Background] Bouffioulx E, Arnould C, Thonnard JL. SATIS-Stroke: A satisfaction measure of activities and participation in the actual environment experienced by patients with chronic stroke. J Rehabil Med. 2008 Nov;40(10):836-43. doi: 10.2340/16501977-0272. PMID 19242621
- [Background] Stucki G. International Classification of Functioning, Disability, and Health (ICF): a promising framework and classification for rehabilitation medicine. Am J Phys Med Rehabil. 2005 Oct;84(10):733-40. doi: 10.1097/01.phm.0000179521.70639.83. No abstract available. PMID 16205428